CLINICAL TRIAL: NCT05183386
Title: Histological Outcome of the Use of Different Biomaterials for Fresh Socket. A Split Mouth Design
Brief Title: Histological Outcome of the Use of Different Biomaterials for Fresh Socket Regeneration. A Split-mouth Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Professor in Prosthodontics, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SocketRegenerationExp
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The dental socket heals spontaneously
- Experimental group (Experimental): Distinct bone graft regeneration strategies (PRGF, Autologous bone and DFDBA)
  Interventions: Procedure: dental socket regeneration

INTERVENTIONS:
Procedure: dental socket regeneration — after a dental extraction the fresh socket is filled with graft materials and compared with the spontaneous healing (control)
  Arms: Experimental group

SUMMARY:
Purpose: The aim of this study was to analyze the quality of bone regeneration in fresh sockets using four different materials and at different times points.

Materials and Methods: A split-mouth clinical trial was designed to evaluate the histological and histomorphometrical characteristics of fresh sockets from 30 patients. One socket per patient will healed spontaneously (control) and, at least, one fresh socket, will be grafted with platelet-rich growth factor (PRGF), PRGF+autologous bone, autologous bone or PRGF+demineralized freeze dried bone allograft (DFDBA). The day of the implant placement, biopsies will be taken at different time points divided into three assessment groups: short duration (2-4 months), intermediate duration (5-6 months) and long duration (7-12 months). The histologic findings will be assessed to quantify the trabeculae pattern, the degree of mineralization and the quality of bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of at least one bilateral tooth extraction due to one or more of the following causes:

  * periodontal disease,
  * vertical fracture
  * included teeth.
* Patients seeking dental implant to replace their missing teeth.
* All sockets should have intact or partially conserved buccal wall according to Elian´s classification (Type I, II).

Exclusion Criteria:

* Patients under 18 years old.
* Patients with a severely untreated periodontal disease.
* Smokers of more than 15 cigarettes a day.
* patients suffering from any systemic disease requiring pharmacological treatment.
* Patients whose socket´s buccal wall is totally missing after tooth extraction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Degree of mineralization | 2-12 months
  Histological Assessment by Von Kossa Stain of the degree of the mineralization in the regenerated bone inside the alveolar walls
type of bone maturation | 2-12 months
  Histological Assessment by Goldner Trichromic Stain of the grade of maturation in the regenerated bone inside the alveolar walls